CLINICAL TRIAL: NCT01565395
Title: Randomized Double Blind Placebo Controlled Cross-Over Study of Incobotulinum Toxin A (Xeomin®) for Troublesome Sialorrhea in Parkinson's Disease (PD)/Parkinsonism and Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Incobotulinum Toxin A for Sialorrhea in Parkinson's Disease (PD)/Parkinsonism and Amyotrophic Lateral Sclerosis (ALS)
Acronym: Xeomin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not recruit ALS participants, hence ALS arm discontinued
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Merz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Pushpa Narayanaswami, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011P000304
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Parkinson Disease; Amyotrophic Lateral Sclerosis
Keywords: ALS; PD
MeSH Terms: conditions — Parkinson Disease; Amyotrophic Lateral Sclerosis | interventions — incobotulinumtoxinA; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Xeomin Injections (Experimental): Fifteen units (0.15 ml) of incobotulinum toxin A injected into each parotid gland and 20 units (0.2 ml) to each submandibular gland for a total dose of 70 units using anatomical landmarks for ALS Twenty units (0.2ml) injected into each parotid gland and 30 units (0.3 ml) to each submandibular gland for a total dose of 100 units using anatomical landmarks for PD/parkinsonism
  Interventions: Drug: Incobotulinum Toxin A
- Placebo (Placebo Comparator): 0.15 ml sterile 0.9% saline injected into each parotid gland and 0.2 ml to each submandibular gland using anatomical landmarks for ALS 0.2ml injected into each parotid gland and 0.3 ml to each submandibular gland using anatomical landmarks for PD/parkinsonism
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Incobotulinum Toxin A — Xeomin 70-100 units injected in the parotid and submandibular glands of subjects
  Other Names: Xeomin
  Arms: Xeomin Injections
Drug: placebo — Sterile preservative free 0.9% saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Incobotulinum Toxin A (Xeomin®) injections into the parotid and submandibular glands in patients with Parkinson's Disease/Parkinsonism and Amyotrophic Lateral Sclerosis (ALS) with troublesome sialorrhea.

DETAILED DESCRIPTION:
Participants will be recruited if they have Parkinson's disease, Parkinsonism. Inclusion and exclusion criteria are summarized below. Participants will be screened at the first visit to make sure they are eligible for the trial. They will then undergo baseline testing including neurologic evaluation, questions to assess their memory and cognitive status and evaluation of their disease status using parts of the Unified Parkinsons's Disease Ratings Scale (UPDRS) that are routinely used to follow disease progression. They will be given a questionnaire to evaluate the severity of their drooling. Their saliva production will be measured by having them spit into a cup for 5 minutes, twice.

At the first visit, after making sure they are eligible for the study and performing the baseline testing and procedures, they will be given either Xeomin or placebo (saline injections without medication) injections in the 4 glands that produce saliva. They will not know which injection they received. This visit will take about 2 hours. They will be followed up every month and asked about side effects, have neurologic evaluation and ALS-FRS testing and fill-in the questionnaire for drooling severity. Saliva volume will be measured as done at the first visit. At either Month 4 or 5, participants will receive the second injection. This will be a "cross-over" injection, i.e., if they received Xeomin at the first injection they will receive saline at the second and vice versa. Thus, all participants will receive the study medication Xeomin, either as the first injection or the second injection at 4 months or 5 months. The follow up after the second injection will be one monthly visit for 3 months, with similar evaluations as described above. The follow-up visit will take about 1 hour each.

ELIGIBILITY:
Inclusion Criteria: Hypothesis: Xeomin® injections into the parotid and submandibular glands are safe and effective in the treatment of troublesome sialorrhea in patients with PD/Parkinsonism and ALS.

Inclusion criteria are as follows:

For ALS: 1. Patients diagnosed with ALS by el-Escorial Criteria, ages 20-80 with troublesome sialorrhea as defined below**.

For PD/ Parkinsonism: 1. PD, Multiple Systems Atrophy (MSA), or Progressive Supranuclear Palsy (PSP) diagnosed by clinical criteria, ages 20-80 with troublesome sialorrhea as defined below**.

**Troublesome sialorrhea is defined as grade 3 or more (grade 3 is marked excess of saliva with some drooling) or more on the UPDRS Part 2 Sialorrhea grading scale:[33] (Appendix 1)

For both groups:

1. Swallowing function: FOIS scale* 5 or greater (see appendix 1 for scale)
2. If patients have been treated with other medications for sialorrhea earlier, they should be off the medications at least 4 weeks prior to the baseline evaluation.
3. If they are on other medications for sialorrhea at the time of the baseline evaluation, the doses will be held stable throughout the period of the study.
4. Women of child bearing age will need to be on a reliable method of birth control for the duration of the study.

Exclusion criteria

For both PD and ALS:

1. Current use of Coumadin
2. Concurrent significant medical illness.
3. History of myasthenia gravis or Lambert-Eaton Syndrome
4. Ongoing substance abuse
5. History of unreliable follow-up
6. Past use of Xeomin® or other botulinum toxin preparations
7. Cognitive impairment, defined as a score ≤ 23/30 on the Mini Mental Status Exam.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in objectively measured salivary volume between baseline and one month post-injection in the Xeomin group as compared to placebo | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Pushpa Narayanaswami, ME, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No